CLINICAL TRIAL: NCT07093203
Title: Pharmacokinetic of Rezafungin in the Plasma and the Peritoneal Fluid of Critically Ill Patients With Intra-abdominal Candidiasis Requiring Abdominal Surgery
Brief Title: Rezafungin Peritoneal Diffusion for Intra-abdominal Candidiasis
Acronym: REAREZ
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024PI230
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-06

CONDITIONS: Intra-Abdominal Infection; Candida; Abdominal Surgery Patients; Critically Ill Intensive Care Unit Patients
Keywords: candida; intra-abdominal candidiasis; abdominal surgery; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Intraabdominal Infections; Torulopsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult critically ill patients with suspected or confirmed intra-abdominal candidiasis

SUMMARY:
ntra-abdominal candidiasis is a serious infection common in critically ill patients, often leading to high mortality if not treated quickly. Standard antifungal treatments may be less effective due to growing resistance and poor drug penetration into the abdominal cavity. In critically ill patients, drug levels can vary widely due to factors like surgery, inflammation, fluid resuscitation, or extracorporeal support, increasing the risk of underdosing. Rezafungin is a new antifungal agent with a long half-life and broad activity against Candida species, offering potential advantages in this setting. However, there is currently no data on its concentration or effectiveness in the peritoneal fluid of patients with intra-abdominal sepsis. Its long half-life, coupled with repeated pharmacokinetic variations in critical care settings and the risk of insufficient concentrations, may hinder its use in this population.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* with a suspected intra-abdominal candidiasis requiring abdominal surgery
* and receiving the administration of rezafungin as first-line empirical antifungal treatment just before the abdominal surgery
* and having abdominal drain for at least 2 days after the surgery

Exclusion Criteria:

* death expected within 24h
* decline to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective PK study of critically ill adult patients with proven or suspected intra-abdominal candidiasis who are admitted to the surgical ICU at the university hospital of Nancy (France).
  Adult critically ill patients with suspected intra-abdominal candidiasis requiring abdominal surgery and administration of rezafungin as first-line empirical antifungal treatment just before the abdominal surgery, abdominal drain for at least 2 days after the surgery.
  Intra-abdominal candidiasis is defined following the 2024 consensus of FUNDICU
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Peritoneal/Plasma Penetration Ratio of Rezafungin | From 0 to 3 hours after rezafungin administration
  Penetration ratio of rezafungin will be calculated as the ratio of the area under the concentration-time curve from 0 to 3 hours (AUC₀-₃h) in peritoneal fluid compared to plasma in critically ill patients undergoing abdominal surgery for suspected or proven intra-abdominal candidiasis

SECONDARY OUTCOMES:
Plasma Concentration-Time Profile of Rezafungin | From 0 to 168 hours after the first rezafungin administration
  Area under the concentration-time curve (AUC) of rezafungin in plasma will be calculated over three time intervals: AUC₀-₂₄h, AUC₀-₄₈h, and AUC₀-₁₆₈h to describe the evolution of plasma concentrations during treatment
Peritoneal Concentration-Time Profile of Rezafungin | From 0 to 48 hours after the first rezafungin administration
  Area under the concentration-time curve (AUC) of rezafungin in peritoneal fluid will be calculated over two time intervals: AUC₀-₂₄h and AUC₀-₄₈h to describe the evolution of peritoneal concentrations during treatment.
Target Attainment in Peritoneal Fluid at the Time of Surgery | At the time of abdominal surgery (within the first 3 hours after rezafungin administration)
  Proportion of patients achieving the pharmacodynamic target in peritoneal fluid, defined as AUC₀-₃h / MIC > 40, measured at the time of surgery.
Postoperative Target Attainment in Plasma | From 0 to 168 hours after the first rezafungin administration
  Proportion of patients achieving the pharmacodynamic target in plasma, defined as AUC₀-₁₆₈h / MIC > 40
Factors Associated with Target Attainment in Peritoneal Fluid | From 0 to 48 hours after the first rezafungin administration
  Analysis of clinical and biological covariates associated with pharmacokinetic variability and the achievement of pharmacodynamic targets in peritoneal fluid
Association Between Pharmacodynamic Target Attainment and Day-28 In-Hospital Mortality | From rezafungin administration to Day 28 post-treatment
  Comparison of Day-28 in-hospital mortality rates between patients who did and did not achieve pharmacodynamic targets in plasma and/or peritoneal fluid

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: Undecided